CLINICAL TRIAL: NCT06974409
Title: The Effects of Foam Rolling on Double-leg Squat Force Distribution
Brief Title: This Study Will Compare Force Production in Double-leg Squats of College Students Before and After a Standardized Foam Rolling Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Redlands (Other)
Responsible Party: Principal Investigator, Kendra Nelson, Doctor, University of Redlands
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Protocol #2025-003-Redlands
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Force Production; Pain Intensity Assessment

STUDY DESIGN:
Intervention Model Description: Single Group Assessment .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foam Rolling Regime (Experimental): 2-minute quadriceps foam rolling regime
  Interventions: Device: foam roller

INTERVENTIONS:
Device: foam roller — foam rollers with grids, knobs, and spikes

SUMMARY:
This study is a within-subject controlled trial . The investigators will compare unilateral force production in a bodyweight double-leg squat before and after a standardized foam rolling session with the use of Vald ForceDecks. TheForceDecks use sensors embedded within separate plates to record the forces exerted. Participants will have their weight, height, and dorsiflexion range of motion measured prior to performing 3 double-leg squats. Participants will then be instructed on the foam rolling technique. They will perform the technique on each quadriceps group and will state their pain level at 30 seconds and at 2 minutes using the VAS pain scale.

DETAILED DESCRIPTION:
The invetigators will compare independent bilateral double-leg squat force productions before and after a structured foam rolling routine. Participants will first be measured for height, weight, and dorsiflexion ROM (SADS; standing ankle dorsiflexion screen). Quadriceps muscle belly length will be determined by measuring from the ASIS to the superior pole of the patella and marking the middle 2/3 of the region. Participants will then stand on VALD ForceDecks for normalization. (The ForceDecks use sensors embedded within separate plates to record the forces exerted by each leg.) With hands on hips, participants will perform three body weight double leg squats (squatting above 90 degrees of knee flexion). Participants will then watch a demonstration of single leg quadriceps foam rolling which will consist of 3-point contact in a plank position with the targeted leg not having contact with the ground. Participants will be cued for continuous motion on a count of 3 seconds in each direction without pausing. Participants will be asked to respond to a visual analog scale for pain at 30 seconds and at 2 minutes (end of session). Participants will be given a 30-second rest between sides. Upon completion, participants will return to the ForceDecks and perform 3 additional body weight double-leg squats with hands on hips (approximate same depth of squat as the initial set).

ELIGIBILITY:
Inclusion Criteria: university student; 18-22 years of age -

Exclusion Criteria: unable to get up from the ground without assistance; current lower extremity injury; prior lower extremity surgery in the past 10 years

-

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Force Production | 30 minutes
  Unilateral lower extremity force production during a single-leg squat.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Redlands, Redlands, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be used for this particular study.

REFERENCES:
- [Background] Hendricks S, Hill H, Hollander SD, Lombard W, Parker R. Effects of foam rolling on performance and recovery: A systematic review of the literature to guide practitioners on the use of foam rolling. J Bodyw Mov Ther. 2020 Apr;24(2):151-174. doi: 10.1016/j.jbmt.2019.10.019. Epub 2019 Nov 2. PMID 32507141
- [Background] Plisky PJ, Bullock GS, Garner MB, Ricard R, Hayden J, Huebner B, Schwartzkopf-Phifer K, Kiesel K. The Dorsiflexion Range of Motion Screen: A Validation Study. Int J Sports Phys Ther. 2021 Apr 1;16(2):306-311. doi: 10.26603/001c.21253. PMID 33842026
- [Background] Pardo E, El Behi H, Boizeau P, Verdonk F, Alberti C, Lescot T. Reliability of ultrasound measurements of quadriceps muscle thickness in critically ill patients. BMC Anesthesiol. 2018 Dec 27;18(1):205. doi: 10.1186/s12871-018-0647-9. PMID 30591032
- [Background] Michalak B, Kopiczko A, Gajda R, Adamczyk JG. Recovery effect of self-myofascial release treatment using different type of a foam rollers. Sci Rep. 2024 Jul 9;14(1):15762. doi: 10.1038/s41598-024-66577-x. PMID 38982124
- [Background] Junker D, Stoggl T. The Training Effects of Foam Rolling on Core Strength Endurance, Balance, Muscle Performance and Range of Motion: A Randomized Controlled Trial. J Sports Sci Med. 2019 Jun 1;18(2):229-238. eCollection 2019 Jun. PMID 31191092
- [Background] Healey KC, Hatfield DL, Blanpied P, Dorfman LR, Riebe D. The effects of myofascial release with foam rolling on performance. J Strength Cond Res. 2014 Jan;28(1):61-8. doi: 10.1519/JSC.0b013e3182956569. PMID 23588488